CLINICAL TRIAL: NCT02861222
Title: Myocet® in Children With Relapsed or Refractory Non-brainstem Malignant Glioma
Acronym: MYOCET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-017803-27
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MYOCET (Experimental): 2 treatments of doxorubicin are administered at 60 mg/m²/day or 75 mg/m²/day in single dose in 1-hour perfusion each 21 days. A maximum of 6 treatments/patient is administered.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin
  Other Names: MYOCET

SUMMARY:
The purpose of this study is to determine the toxicity and tolerance of Myocet® in children and adolescents with refractory or relapsed malignant glioma, with a dose diminished of 20% of the dose recommended for adults and a dose recommended for adults, administered in single dose in 1-hour perfusion each 21 days.

Other purposes are to determine the recommended dose of Myocet and to assess the response to drug. Pharmacokinetics of doxorubicin (free and encapsulated forms) and its metabolite doxorubicinol during 72 hours after Myocet administration will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients having received at least one cycle of chemotherapy after radiotherapy
* Patients having grade III or IV (WHO) glioma, not localized in brainstem
* Tumor measurable with magnetic resonance imaging
* Absence of other concomitant anti-cancer treatments
* Absence of chemotherapy for 4 weeks; 6 weeks if nitrosourea
* Good general health and nutritional status according to NCI-CTC scale (version 3) (appendix 6)
* Lansky score > 50% or Karnofsky > 50 in children older than 12 years
* Absence of organ toxicity (grade > 2 according to NCI-CTC criteria (version 3)
* Hematology: polynuclear neutrophil count > 1.0 x 109/l
* Hematology: platelet count > 100 x 109/l
* Liver function: bilirubinemia < 1.5 normal value
* Liver function: ASAT and ALAT levels < 2.5 normal values
* Liver function: prothrombin level > 70%
* Liver function: fibrinogen > 1.5 g/l
* Renal function: creatinemia < 1.5 normal value/age
* Cardiac function: EF > 60% and/or SF > 30%
* Signature of informed consent by patient if adolescent, by 2 parents or legal guardian if minor patient
* For patients with childbearing potential, a contraceptive method is compulsory. This contraception must be continued 6 months after Myocet treatment end
* For patients with childbearing potential, negative pregnancy test (betahCG test)

Exclusion Criteria:

* Non compliance with eligibility criteria
* Severe or life-threatening infection
* Non controlled evolutive or symptomatic intracranial hypertension
* History of Myocet treatment, but patients could be treated with anthracyclines if cardiac function is normal
* Hypersensibility to the active substance, to premixtures or one of excipients
* Pregnancy and breastfeeding

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
General health evaluation | From day 21 post-dose
  NCI-CTC scale, version 3, appendix 6
Changes in neurological condition related to the tumor (motor deficit, sensory deficit, cranial nerves pairs defect, cerebellar syndrome, vertebrobasilar defect, pyramidal tract syndrome) assessed during clinical examination | From day 21 post-dose
Complete blood count (platelet included) | 2 times/week from day 0
ALAT/ASAT measurement | From day 21 post-dose
Bilirubin test | From day 21 post-dose
Prothrombin test | From day 21 post-dose
Fibrin measurement | From day 21 post-dose
Partial thromboplastin time test | From day 21 post-dose
Creatinine blood test | From day 21 post-dose
Analysis of the electrolyte composition of the blood | From day 21 post-dose
Blood urea analysis | From day 21 post-dose
Glycemia analysis | From day 21 post-dose
Calcemia analysis | From day 21 post-dose
Protidaemia analysis | From day 21 post-dose
Normality of ECG | From day 21 post-dose
Echocardiography with analysis of ventricular ejection and shortening fractions | From day 21 post-dose

SECONDARY OUTCOMES:
Measure of initial tumors with MRI | from day 42, after each 2 treatments
Antitumoral activity (radiological criteria of SIOP protocol) | from day 42, after each 2 treatments
Plasma measurement of free doxorubicin | 0, 2, 5, 11, 47, 71 hours after the first dose
Plasma measurement of encapsulated doxorubicin | 0, 2, 5, 11, 47, 71 hours after the first dose
Plasma measurement of doxorubicinol | 0, 2, 5, 11, 47, 71 hours after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Chastagner, Principal Investigator — Service d'Hémato-Oncologie pédiatrique, Hôpital d'Enfants, CHU Nancy
Locations (7):
- France (7):
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CHU, Hôpital d'Enfants de la Timone, Marseille
  - Institut Curie, Paris
  - Unité d'Hémato-Oncologie, CHU, Hôpital des enfants, Toulouse
  - CHU, Hôpital d'Enfants, Vandœuvre-lès-Nancy
  - Institut Gustave-Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No